CLINICAL TRIAL: NCT00882505
Title: Comparison of 25-hydroxy Vitamin D Level in Caucasian Women Receiving Vitamin D Supplementation and Not Receiving Supplementation: a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU8461
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D supplement (Experimental): Receive vitamin D supplements.
  Interventions: Dietary Supplement: vitamin D
- Placebo (Placebo Comparator): Receive placebo pills
  Interventions: Other: Placebo
- Tanning bed user (No Intervention): Regular tanning bed users will be assessed for their vitamin D levels.

INTERVENTIONS:
Dietary Supplement: vitamin D — Subject will receive vitamin d supplements
  Arms: Vitamin D supplement
Other: Placebo — Subject will receive a placebo.
  Arms: Placebo

SUMMARY:
The objective of this study is to assess whether vitamin D supplements are sufficient to increase females who are deficient or borderline deficient in vitamin D levels to normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Caucasian women, ages 18-47
* Subjects in good health
* Tanning bed group: regular tanning bed user at least once a week for previous 10 weeks

Exclusion Criteria:

* Pregnancy and lactation
* Subjects with liver disease, renal disease, multiple myeloma, parathyroid disease, irritable bowel disease, celiac disease, cystic fibrosis and pancreatic disease
* Subjects with hypocholesterolemia and primary hyperparathyroidism
* Subjects taking the following medications:

  * Steroids
  * Orlistat
  * Lipid lowering medication: cholestyramine, statins
  * Antiepileptic drugs: phenobarbital and phenytoin
  * Currently on vitamin D supplements or using any medication contain vitamin D i.e. cod liver oil, topical calcipotriol or history of use within 1 month
  * Rifampicin, isoniazid
  * Ketoconazole
* Subjects currently on UV therapy

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
For the randomized controlled trial, the primary outcome measure is comparison of the change in vitamin D levels in the vitamin D supplementation group and the placebo group. | 3 months
For the comparative study, the primary outcome measure is comparison of the vitamin D level for tanning bed users compared to the level for non-tanning bed users. | 3 months

SECONDARY OUTCOMES:
The secondary outcome measures include evaluation of changes in other laboratory parameters associated with change in vitamin D level. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States